CLINICAL TRIAL: NCT03062254
Title: Metabolic Change in Prostate Cancer Bone Metastases on 68Ga-HBED-CC-PSMA PET/CT Following Radium-223 Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, MD, Chief of Nuclear Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-029
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: PSMA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radium-223 (Experimental)
  Interventions: Drug: radium-223 dichloride

INTERVENTIONS:
Drug: radium-223 dichloride — 6 doses of Radium-223

SUMMARY:
Broadly, the objective of this study is to evaluate the fractional decline of intensity of tracer uptake measured by SUVmax on 68Ga-PSMA PET/CT in bone metastases from prostate cancer following treatment with radium-223 as a surrogate marker for tumor cell killing.

ELIGIBILITY:
Inclusion Criteria

* Resident of Canada
* Male sex
* Age 18 years or older
* Progressive (symptoms, conventional imaging, PSA, bone scan, FCH PET/CT or other) castration-resistant prostate cancer in the judgment of the treating physician without change in systemic anti-neoplastic therapy since documented progression
* Six or greater bone metastases robustly-avid on recent (4 weeks) MDP or NaF scintigraphy
* Recently failed (within 3 months) or failing novel androgen receptor pathway inhibitors (abiraterone + prednisone or enzalutamide) with intention of continuing the drug for at least 7 months OR minimum 14 day washout period from either agent prior to study enrollment
* No known visceral metastases or adenopathy greater than 3 cm short axis on conventional imaging
* Not received docetaxel for castration-resistant disease
* ECOG performance status 0 - 2, inclusive
* Life expectancy of greater than 6 months
* Serum testosterone less than or equal to 50 ng/dl
* Hemoglobin greater than or equal to 100 g/L with no blood transfusions or EPO in preceding 3 weeks
* Neutrophils greater than or equal to 1.5 x109/L
* Platelets greater than or equal to 100 x109/L
* No prior hemi-body radiotherapy
* No impending or established spinal cord compression
* No unmanageable fecal incontinence
* Patient has good IV access
* Able to understand and provide written informed consent

Exclusion Criteria

* Planned change in systemic anti-neoplastic therapy during the approximately 7 month trial
* Unable to tolerate the physical/logistical requirements of a PET/CT scan including lying supine for up to 30 minutes with the arms above the head and tolerating intravenous cannulation for injection of the study drug.
* Medically unstable patients (e.g. acute cardiac or respiratory distress or hypotensive, etc.)
* Patients who exceed the safe weight limit of the PET/CT bed (approximately 400 lbs.) or who cannot fit through the PET/CT bore (70 cm diameter)
* Patients who are claustrophobic

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male only
Enrollment: 14 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
SUV-max | 6 months
  fractional decline of intensity of tracer uptake measured by SUVmax on 68Ga-PSMA PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided